CLINICAL TRIAL: NCT01288768
Title: Is a Knee Arthroscopy of Any Benefit for the Middleaged Patient With Meniscal Symptoms?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Hakan Gauffin, MD PhD, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/6-31
Record Dates: First submitted 2011-01-26; First posted 2011-02-02 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Meniscus Injury
Keywords: Meniscal injury; Knee arthroscopy; Middleaged; Functional outcome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthroscopy (Active Comparator): Knee arthroscopy + Exercise therapy
  Interventions: Procedure: Knee arthroscopy
- Exercise therapy (No Intervention): Exercise therapy alone

INTERVENTIONS:
Procedure: Knee arthroscopy — Knee arthroscopy within 4 weeks.
  Arms: Arthroscopy

SUMMARY:
The purpose of this study is to determine whether a knee arthroscopy is effective in the treatment of middleaged patients with meniscal symptoms also receiving a standardised exercise program.

DETAILED DESCRIPTION:
There are no studies proving a significant positive effect of a knee arthroscopy in middleaged patients with meniscal symptoms in excess of a structured rehabilitation program. In this study consecutive patients aged 45-64 years referred to the orthopaedic department at the University hospital Linköping for a suspected meniscal injury will be randomised to a rehabilitation program or a knee arthroscopy + the same rehabilitation program. Functional tests will be performed by a physiotherapist. There will be patient administrated questionaries sent out after 3 and 12 month.

ELIGIBILITY:
Inclusion Criteria:

* All (consecutive) patients referred to the orthopaedic department in Linköping for a suspected meniscal injury
* Age:45-64 years old
* No gonarthrosis (Ahlbäck=0) on standing radiographs

Exclusion Criteria:

* Rheumatic disease
* Patellofemoral arthrosis
* Fibromyalgia
* A knee or hip replacement
* A neurologic disorder including stroke
* A contraindication for an operation
* Catching or locking for more than 2 seconds more than once a week
* A permanent extension deficit
* Patients who cannot understand instructions in Swedish

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2010-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
KOOS (Knee injury and Osteoarthritis Outcome Score); Pain subscale | 12 month
  KOOS is a 42 item selfadministrated questionnaire with 5 separate subscales; pain, symptoms, activities of daily living (ADL), sport and recreation, quality of life (QoL). A change of approximately 10 is considered a clinical important difference (CID). At 12 month after the randomization the "arthroscopy+exercise therapy" arm will be compared to the "exercise therapy alone" arm.

SECONDARY OUTCOMES:
KOOS (Knee injury and Osteoarthritis Outcome Score) | 3 month
Tegner activity scale | 12 month
KOOS (Symptoms, ADL, Sport/rec, QOL subscores) | 12 month
Functional tests | 3 month
  Squatting (possible without pain, possible with pain, not possible). SOLEC ( one-legged stance) barefoot. Best time for three trials. Standing up from a chair on one leg, maximum repetitions in 30 sec. All test supervised by a physiotherapist.

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Gauffin, MD PhD, Principal Investigator — Orthopaedic dept. University Hospital, Linköping, Sweden.
Locations (1):
- Orthopaedic dept. University Hospital Linköping, Linköping, Sweden

REFERENCES:
- [Background] Englund M, Roos EM, Roos HP, Lohmander LS. Patient-relevant outcomes fourteen years after meniscectomy: influence of type of meniscal tear and size of resection. Rheumatology (Oxford). 2001 Jun;40(6):631-9. doi: 10.1093/rheumatology/40.6.631. PMID 11426019
- [Background] Englund M, Guermazi A, Gale D, Hunter DJ, Aliabadi P, Clancy M, Felson DT. Incidental meniscal findings on knee MRI in middle-aged and elderly persons. N Engl J Med. 2008 Sep 11;359(11):1108-15. doi: 10.1056/NEJMoa0800777. PMID 18784100
- [Background] Ericsson YB, Dahlberg LE, Roos EM. Effects of functional exercise training on performance and muscle strength after meniscectomy: a randomized trial. Scand J Med Sci Sports. 2009 Apr;19(2):156-65. doi: 10.1111/j.1600-0838.2008.00794.x. Epub 2008 Apr 6. PMID 18397193
- [Background] Herrlin S, Hallander M, Wange P, Weidenhielm L, Werner S. Arthroscopic or conservative treatment of degenerative medial meniscal tears: a prospective randomised trial. Knee Surg Sports Traumatol Arthrosc. 2007 Apr;15(4):393-401. doi: 10.1007/s00167-006-0243-2. Epub 2007 Jan 10. PMID 17216272
- [Background] Larsson AC, Petersson I, Ekdahl C. Functional capacity and early radiographic osteoarthritis in middle-aged people with chronic knee pain. Physiother Res Int. 1998;3(3):153-63. doi: 10.1002/pri.137. PMID 9782518
- [Background] Paradowski PT, Englund M, Roos EM, Lohmander LS. Similar group mean scores, but large individual variations, in patient-relevant outcomes over 2 years in meniscectomized subjects with and without radiographic knee osteoarthritis. Health Qual Life Outcomes. 2004 Jul 27;2:38. doi: 10.1186/1477-7525-2-38. PMID 15279676
- [Background] Roos EM, Roos HP, Ekdahl C, Lohmander LS. Knee injury and Osteoarthritis Outcome Score (KOOS)--validation of a Swedish version. Scand J Med Sci Sports. 1998 Dec;8(6):439-48. doi: 10.1111/j.1600-0838.1998.tb00465.x. PMID 9863983
- [Background] Roos EM, Roos HP, Ryd L, Lohmander LS. Substantial disability 3 months after arthroscopic partial meniscectomy: A prospective study of patient-relevant outcomes. Arthroscopy. 2000 Sep;16(6):619-26. doi: 10.1053/jars.2000.4818. PMID 10976123
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Roos EM, Bremander AB, Englund M, Lohmander LS. Change in self-reported outcomes and objective physical function over 7 years in middle-aged subjects with or at high risk of knee osteoarthritis. Ann Rheum Dis. 2008 Apr;67(4):505-10. doi: 10.1136/ard.2007.074088. Epub 2007 Aug 17. PMID 17704069
- [Background] Tegner Y, Lysholm J. Rating systems in the evaluation of knee ligament injuries. Clin Orthop Relat Res. 1985 Sep;(198):43-9. PMID 4028566
- [Background] Wood L, Peat G, Thomas E, Hay EM, Sim J. Associations between physical examination and self-reported physical function in older community-dwelling adults with knee pain. Phys Ther. 2008 Jan;88(1):33-42. doi: 10.2522/ptj.20060372. Epub 2007 Nov 20. PMID 18029391
- [Derived] Sonesson S, Springer I, Yakob J, Hedevik H, Gauffin H, Kvist J. Knee Arthroscopic Surgery in Middle-Aged Patients With Meniscal Symptoms: A 10-Year Follow-up of a Prospective, Randomized Controlled Trial. Am J Sports Med. 2024 Jul;52(9):2250-2259. doi: 10.1177/03635465241255653. PMID 39101738
- [Derived] Sonesson S, Kvist J, Yakob J, Hedevik H, Gauffin H. Knee Arthroscopic Surgery in Middle-Aged Patients With Meniscal Symptoms: A 5-Year Follow-up of a Prospective, Randomized Study. Orthop J Sports Med. 2020 Jan 27;8(1):2325967119893920. doi: 10.1177/2325967119893920. eCollection 2020 Jan. PMID 32047825
- [Derived] Gauffin H, Sonesson S, Meunier A, Magnusson H, Kvist J. Knee Arthroscopic Surgery in Middle-Aged Patients With Meniscal Symptoms: A 3-Year Follow-up of a Prospective, Randomized Study. Am J Sports Med. 2017 Jul;45(9):2077-2084. doi: 10.1177/0363546517701431. Epub 2017 Apr 21. PMID 28429967
- [Derived] Gauffin H, Tagesson S, Meunier A, Magnusson H, Kvist J. Knee arthroscopic surgery is beneficial to middle-aged patients with meniscal symptoms: a prospective, randomised, single-blinded study. Osteoarthritis Cartilage. 2014 Nov;22(11):1808-16. doi: 10.1016/j.joca.2014.07.017. Epub 2014 Jul 30. PMID 25086401